CLINICAL TRIAL: NCT06174480
Title: Evaluation of the Response to Hypoxia at Rest and During Exercise in a Healthy Subject After a Cryostimulation Exposure
Acronym: CRYOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Poitiers University Hospital (Other)
Collaborators: Poitiers University - Laboratoire MOVE UR 20296, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CRYOX
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-12

CONDITIONS: Hypoxia; Cryostimulation; Metabolism; Autonomic Nervous System; Exercise; Adaptation
MeSH Terms: conditions — Hypoxia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants will not undergo cryostimulation exposure but will only receive 2 1-hour hypoxia sessions at FiO2 13.5% for 1 hour, at 2-week interval
- Cryostimulation Group (Experimental): Participants will be exposed to cryostimulation (-50°C, forced ventilation for 3 minutes) during 20 sessions over 2 weeks and will undergo 2 hypoxia sessions at FiO2 13.5% for 1 hour, at 2-week interval
  Interventions: Other: Cryostimulation

INTERVENTIONS:
Other: Cryostimulation — Cryostimulation (-50°C, forced ventilation for 3 minutes) during 20 sessions over 2 weeks.
  Arms: Cryostimulation Group

SUMMARY:
Many information is available regarding human adaptations to cold or hypoxia. Adaptations to these environments and physical exercise constitute responses to physiological stress aimed at amplifying the organism's reactions and improving its performance. However, studies conducted so far to understand these adaptations and their underlying mechanisms have been organized in a dissociated manner, with each study focusing on only one of these specific situations (cold, hypoxia, or exercise). Understanding cross-adaptations is crucial, as human beings are often simultaneously exposed to several of these stimuli, and understanding this cross-exposure can be considered a prerequisite for pre-acclimatization strategies to these different environments.

Cross-adaptations has been defined as follows: "It simply involves considering that long-term exposure (either continuous or intermittent) to a given unfavorable environment not only increases tolerance to that particular environment but also leads to gains or losses of tolerance to other unfavorable factors that the adapted organism had never encountered before." When specifically examining cross-adaptations to cold and hypoxia, only one study focusing on the human model is available. The lack of perspectives and positions regarding the results calls for further investigations.

The main objective of this study is to assess the effect of repeated exposures to cryostimulation on the variation of the respiratory exchange ratio in hypoxia during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Having a high level of physical activity according to the criteria of the World Health Organization, assessed using the Global Physical Activity Questionnaire (GPAQ);
* No exposure to cryostimulation or hypoxia (FiO2 13.5%, equivalent to an altitude of 3500 m) in the last 90 days;
* No planned sports competition during the 4 weeks of the protocol;
* Maintaining a stable physical activity level (regular training, without interruption or specific competition, including sports training programs) anticipated for 4 weeks;
* No history of respiratory conditions (asthma, respiratory allergies, exercise-induced asthma, exertional dyspnea);
* Absence of any chronic medical condition;
* No ongoing medication treatments;
* Covered by a French Social Security;
* Informed consent, signed by the subject after clear and fair information about the study.

Exclusion Criteria:

* Subject under treatment;
* Simultaneous participation in another clinical research study;
* Individuals with enhanced protection, namely minors, individuals deprived of liberty by judicial or administrative decision, persons staying in a healthcare or social facility, adults under legal protection, and finally, patients in emergency situations;
* Subject presenting a contraindication to hypoxia and/or cryostimulation.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
variation of the respiratory quotient during exercise | Comparing the average values obtained during exercise in hypoxia at baseline and after 15 days.
  respiratory exchange ratio will be measured continuously using a portable metabolic station to analyze gas exchanges

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Laboratoire MOVE UR 20296 - Poitiers University, Poitiers
  - Clinical Investigation Centre INSERM CIC1402 - Poitiers University - CHU POITIERS, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided